CLINICAL TRIAL: NCT02151799
Title: Body Contouring - the Analysis of Non-invasive and Invasive Methods and Their Interventional Effects on Quality of Life
Brief Title: The Effects of Body Contouring: Abdominoplasty and Liposuction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R09166
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Subcutaneous Abdominal Fat; Abdominal Skin Elasticity; Rectus Muscle Diastasis; Unpleasant Body Contour
MeSH Terms: interventions — Abdominoplasty; Lipectomy

ARMS (1):
- Body contouring surgery (Experimental)
  Interventions: Procedure: Abdominoplasty and liposuction

INTERVENTIONS:
Procedure: Abdominoplasty and liposuction

SUMMARY:
The data regarding the effects of aesthetic body contouring is insufficient. Poor results may related to preoperative psychological distress. Studies regarding eating disorder symptoms are lacking. Therefore studies using standardized and validated are needed. We decided to prospectively study quality of life, psychological distress, and eating disorder symptoms in body contouring (abdominoplasty or liposuction) patient populations. Used questionnaires are 15D quality of life, Raitasalo's modification of the Beck Inventory, and the Eating Disorder Inventory. We hypothesize that aesthetic body contouring plastic surgery has notable quality of life effects.

ELIGIBILITY:
Inclusion Criteria:

* patients requesting body contouring surgery

Exclusion Criteria:

* previous abdominal aesthetic surgery, simultaneous other aesthetic surgery at the same time

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2010-01; Primary Completion 2014-02 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Quality of life | 6 months
  15D quality of life questionnaire RBDI mood questionnaire Eating Disorder Inventory questionnaire

REFERENCES:
- [Derived] Saariniemi KM, Salmi AM, Peltoniemi HH, Helle MH, Charpentier P, Kuokkanen HO. Abdominoplasty improves quality of life, psychological distress, and eating disorder symptoms: a prospective study. Plast Surg Int. 2014;2014:197232. doi: 10.1155/2014/197232. Epub 2014 Nov 24. PMID 25506426
- See also: Related Info — http://journals.lww.com/prsgo/Citation/2015/07000/Does_Liposuction_Improve_Body_Image_and_Symptoms.7.aspx